CLINICAL TRIAL: NCT06781684
Title: Ulnar Shaft Fracture Fixation by Antegrade Versus Retrograde Intramedullary k Wires in Children;A Comparative Study
Brief Title: Ulnar Shaft Fracture Fixation by Antegrade Versus Retrograde Intramedullary k Wires in Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Ali, Orthopedic Resident at sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-12-01MS
Record Dates: First submitted 2024-12-31; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Fracture of Ulna Shaft
Keywords: Fixation of pediatric ulna shaft fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antegrade intramedullary k wire group (Active Comparator): k wire entry point is from the olecranon towards the hand before the distal ulnar styloid
  Interventions: Procedure: ulna shaft fracture fixation in children by intramedullary k wire
- Retrograde intramedullary k wire group (Active Comparator): k wire entry point is from the distal ulnar styloid towards the olecranon
  Interventions: Procedure: ulna shaft fracture fixation in children by intramedullary k wire

INTERVENTIONS:
Procedure: ulna shaft fracture fixation in children by intramedullary k wire — * In the 1st group The Antegrade intramedullary k wire with appropriate diameter according to the child ulna diameter is introduced from the olecranon of the fractured ulna,cross the fracture site after good reduction under C arm in the anterioposterior and lateral views and the wire continues until reaching before the distal ulna .
  * In the 2nd group The Retrograde intramedullary k wire with appropriate diameter is introduced from the diatal end of the ulna and cross the fracture site after good reduction under C arm and continues until reaching before the olecranon.

SUMMARY:
This study is made to see and evaluate the outcomes of treating and fixing ulnar shaft fracture in children by antegrade versus retrograde intramedullary k wires

DETAILED DESCRIPTION:
This study is made on children with ulnar shaft fracture and treating their fracture by intramedullary k wires ,dividing them into two groups ,one of them the child ulnar fracture is reduced and fixed by intramedullary antegrade k wire and the other group the fracture is reduced and fixed by retrograde k wire ,and compare the functional, clinical and radiological outcomes between the two groups

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patient
* aging from 4 to 15 years old
* diaphyseal ulnar fracture
* either isolated or combined with radius fracture (both bone).

Exclusion Criteria:

* Segmental fractures
* Montaggia variants
* Gelliazzi fracture
* Fractures associated with radial head fracture - Compound fractures
* Fractures with neurovascular affection

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
The duration of complete union of the bone in every group | The evaluation is done at 2,4,6 and 12 weeks and 3 months
  Each patient is evaluated radiologically after fixing the fracture by x-ray AP and lateral views after 2 week ,4 ,6 ,12 weeks and 3 months to see the time each one taking to complete union .
  -Also clinical and functional evaluation of every patient and timing of ability to use his forearm , ability to do supination and pronation of the forearm , flexion and extension of the elbow and wrist , ability to do ulnar deviation at the level of the wrist and degree of pain and apprehension with each movement ,Degree of pain and tenderness in the fracture site and time taking to complete disappearing of pain and tenderness ,degree of stiffness and need to physiotherapy ,these data is collected from each patient at the time of follow up in the outpatient clinic and recorded for everyone in each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt